CLINICAL TRIAL: NCT06952660
Title: A PROSPECTIVE LOW-INTERVENTIONAL PHASE 4 SINGLE ARM STUDY OF OCULAR ASSESSMENTS IN PATIENTS TREATED WITH TIVDAK® IN RECURRENT OR METASTATIC CERVICAL CANCER
Brief Title: Ocular Assessments in Patients Treated With Tivdak® in Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C5721005
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: Uterine Neoplasms; Genital Neoplasms; Female Urogenital Neoplasms; Neoplasms by Site; Neoplasms Uterine; Cervical Diseases; Uterine Diseases; Genital Diseases, Female; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Genital Diseases Uterine Cervical Neoplasms,; Tisotumab vedotin
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Neoplasms by Site; Uterine Cervical Diseases; Uterine Diseases; Genital Diseases, Female; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tisotumab vedotin (Experimental): Participants will receive tisotumab vedotin by IV infusion.
  Interventions: Drug: TIVDAK

INTERVENTIONS:
Drug: TIVDAK — 2 mg/kg once every 3 weeks (Q3W)

SUMMARY:
TIVDAK is used for the treatment of cervical cancer that has come back after chemotherapy. Chemotherapy is a treatment that uses medicines to stop the growth of cancer cells. This is done either by killing the cells or by stopping them from growing. The purpose of this study is to learn about possible side effects of TIVDAK, specially to any side effect that is related to the eye. A side effect is anything a medicine does to your body that is not part of how the medicine treats disease.

* This study is seeking for participants who: Are willing to take all the required eye tests
* Have not received TIVDAK before
* Do not have any active eye issues.

Participants will receive TIVDAK once every 3 weeks as an infusion that will be injected into the vein. Participants will visit an eye care provider at 3 stages:

* before starting the treatment,
* before each of the first 9 infusions
* then monthly for 3 months after they stop taking TIVDAK. Treatment with TIVDAK will continue until it is not working anymore against the participant's cancer.

ELIGIBILITY:
Inclusion criteria:

1. Must have recurrent or metastatic cervical cancer with disease progression on or after chemotherapy
2. Treating physician has determined that treatment with Tivdak is appropriate for the participant according to US Prescribing Information
3. Must sign an informed consent form indicating that the participant understands the purpose and procedures required for the study and are willing to participate
4. Must be willing to undergo repeated ocular assessments as required by the study and regular clinic visits according to local standard practice of the study site
5. Must agree to use effective contraception according to the US Prescribing Information

Exclusion criteria:

1. Active ocular disease at baseline per investigator assessment
2. Previous treatment with Tivdak
3. Previous administration of an investigational drug within 30 days
4. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may, in the investigator'

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-12-13 (Estimated); Study Completion 2028-12-13 (Estimated)

PRIMARY OUTCOMES:
Type, incidence and severity of ocular adverse events (AEs) | 90 days after the last dose of tisotumab vedotin

SECONDARY OUTCOMES:
Time to resolution of ocular AEs | 90 days after the last dose of tisotumab vedotin
Time to onset of ocular AEs | 90 days after the last dose of tisotumab vedotin
Incidence of serious adverse events (SAEs) | 90 days after the last dose of tisotumab vedotin
AEs leading to dose modifications including treatment discontinuation | 90 days after the last dose of tisotumab vedotin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (38):
  - Mount Sinai Comprehensive Cancer Center - Aventura, Aventura, Florida
  - Broward Health Coral Springs, Coral Springs, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Broward Health Imperial Point, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - HCA Mercy Hospital, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center of Florida, Inc, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Orlando Health Orlando Regional Medical Center, Orlando, Florida
  - Orlando Health Winnie Palmer Hospital for Women & Babies, Orlando, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Cancer Institute St Matthews Campus, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - University Medical Center - New Orleans, New Orleans, Louisiana
  - Trials365, LLC, Shreveport, Louisiana
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Willis Knighton Physician Network - Hematology/Oncology, Shreveport, Louisiana
  - Willis Knighton Physician Network/Gynecologic Oncology Associates, Shreveport, Louisiana
  - WK Eye Institute North, Shreveport, Louisiana
  - St. Dominic - Jackson Memorial Hospital, Jackson, Mississippi
  - St. Dominic Gynecologic Oncology, Jackson, Mississippi
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Miami Valley Hospital South, Centerville, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Texas Oncology - Central South, Austin, Texas
  - Texas Oncology - Central South, Harlingen, Texas
  - Texas Oncology - Central South, McAllen, Texas
  - Texas Oncology - Central South, Waco, Texas
  - Texas Oncology - Central South, Weslaco, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - UVA Health Cancer Care Pantops, Charlottesville, Virginia
- Puerto Rico Cancer Specialists Clinical Trials, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5721005